CLINICAL TRIAL: NCT06530628
Title: Evaluation of Olfactory Stimulation of the Appetite of the Elderly in Long-term Care Units by the Diffusion of Culinary Scents : Proof of Concept.
Brief Title: Prospective Study on Appetite Stimulation by Culinary Scents in the Elderly People
Acronym: APPETIT-SENS
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL22_0295
Record Dates: First submitted 2024-07-26; First posted 2024-07-31 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Elderly People Hospitalized
Keywords: Appetite; Undernutrition; Scents; Elderly in long-term care units
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adult patients resident in Pavillon C of the Pierre Garraud Hospital
  Interventions: Behavioral: Adult patients resident in Pavillon C of the Pierre Garraud Hospital

INTERVENTIONS:
Behavioral: Adult patients resident in Pavillon C of the Pierre Garraud Hospital — Adult patients resident in Pavillon C of the Pierre Garraud Hospital, aged over 70, polypathological, with or without undernutrition.
  The intervention involves the diffusion of culinary odors using diffusers in the unit's hallways, 20 minutes before lunch, from Monday to Friday, for a period of three weeks.
  This experiment will be repeated over 18 weeks (6 cycles), alternating meals without olfactory stimulation (cycles 1, 3 and 5) and meals with stimulation (cycles 2, 4 and 6).
  The 3-week rhythm corresponds to the menu cycle proposed by the Unité Centrale de Production Alimentaire (UCPA). Thus, the menu will be the same whether or not it is associated with the diffusion of culinary scents.

SUMMARY:
Undernutrition affects 2 million people in France, including 400,000 elderly people living at home and 270,000 in nursing homes. It leads to increased morbidity, dependency and mortality. For the elderly in institutions, the activity associated with food intake should remain a source of recurrent pleasure; when altered, it leads to anhedonia and sarcopenia, and increases the risk of infection.

A study conducted with Alzheimer's patients has begun to demonstrate that exposing patients to a food odor 15 min before a meal helps restore their appetite and increase food intake.

A common finding among all the research into undernutrition in the elderly is that olfactory deficits, caused by centrally-cooked and then reheated meals with no appetizing smell, affect the pleasure of eating. As we age, our ability to perceive smells diminishes, as they need to be more intense to be perceived. Diminished pleasure in food odors thus plays a role in the onset of anorexia.

The Pierre Garraud Hospital accommodates 305 residents in 9 long-term care units. One of the concerns of the care teams is to prevent undernutrition.

One of the levers of this prevention is to reinforce the diet to increase the quantity and quality of the elderly's nutrition.

While particular attention is paid to the visual quality of the service and to improving the taste of the food on offer at the Hospices Civils de Lyon, the olfactory component is difficult to mobilize with a centralized food preparation process, even after re-heating in the unit.

However, caregivers have observed a marked appetite for meals prepared in the unit during entertainment activities. The diffusion of strong culinary odors was identified as an appetite vector.

This research hypothesis stems from this experience:

"The diffusion of culinary scents before meals can stimulate residents' appetite in order to encourage increased nutritional intake".

Although the elderly often suffer from olfactory loss, they are able to detect odors when presented at higher concentrations. Olfactory stimulation in a population of elderly people, 2/3 of whom have cognitive impairments, represents a real vector for the reminiscence of memories and the cognitive engagement in the act of eating.

The original idea of this study was to compensate for the absence of odors during the reheating of institutional meals, by stimulating appetite through the diffusion of culinary scents.

This would be a first exploratory proof-of-concept study of the benefits of scent diffusion on food intake and its evolution over time.

ELIGIBILITY:
Inclusion Criteria:

* Resident over 70 years, hospitalized in a long-term care unit at the Pierre GARRAUD Hospital in pavillon C on the first floor (Hospices Civils de Lyon).
* Resident able to eat orally in the dining room or in bedroom.
* Resident who are autonomous for eating, with or without deglutition disorders, with or without the prescription of food supplements, whatever the prescribed texture.
* Resident who does not object to participation in the study or resident with a legal protection measure such as guardianship/curatorship who does not object to the resident's participation in the study.

Exclusion Criteria:

* Resident on parenteral or enteral nutrition.
* Resident in end-of-life care.
* Resident participating simultaneously in another research study, of which the aim is to evaluate a drug or non-drug therapy likely to improve nutrition or weight control.

Ages: 70 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Adult patients resident in Pavillon C of the Pierre Garraud Hospital, aged over 70, polypathological, with or without undernutrition.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2024-12-23 (Actual); Primary Completion 2025-05-16 (Actual); Study Completion 2025-05-16 (Actual)

PRIMARY OUTCOMES:
Food intake of each resident : difference between weights served and weights of food leftovers. It will be compared between periods with olfactory stimulation and periods without. | During the intervention. This experiment will be repeated over 18 weeks (6 cycles), alternating meals without olfactory stimulation (cycles 1, 3 and 5) and meals with stimulation (cycles 2, 4 and 6).
  Every day at lunchtime, the food will be weighed : once before the resident is served, and again when the tray is cleared.

CONTACTS AND LOCATIONS:
Locations (1):
- Pavillon C Hôpital Pierre Garraud / Groupement Hospitalier Nord - HCL, Lyon, France

IPD SHARING:
Plan to Share IPD: No